CLINICAL TRIAL: NCT03226600
Title: A COMPARATIVE STUDY OF ROOT COVERAGE USING OrACELL™ VERSUS SUBEPITHELIAL CONNECTIVE TISSUE GRAFT: A RANDOMIZED CONTROLLED TRIAL
Brief Title: OrACELL™ vs. Connective Tissue in Miller Class 3 Defects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas A&M University (Other)
Collaborators: LifeNet Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2014-0833-BCD-FB
Record Dates: First submitted 2017-05-31; First posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-05

CONDITIONS: Gingival Recession
Keywords: Gingival Recession; Connective Tissue Graft; OrACELL; Decellularized Dermis; Periodontics
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial between two treatment modalities for gingival recession with 6 month follow-up
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Connective Tissue Graft (Active Comparator): Connective Tissue is harvested from the palate of the subject then placed over the recession defect on the facial of the designated tooth. A coronally advanced flap is raised to cover the connective tissue graft and the recession.
  Interventions: Device: Connective Tissue Graft
- OrACELL (Experimental): Allograft Tissue (human dermis) is removed from packing and placed over the recession defect on the facial of the designated tooth. A coronally advanced flap is raised to cover the OrACELL graft and the recession.
  Interventions: Device: OrACELL

INTERVENTIONS:
Device: OrACELL — OrACELL is human dermis that undergoes the MATRACELL process. MATRACELL is a patented and validated process that renders allograft tissue acellular, without compromising the biomechanical or desired biochemical properties of an allograft bio-implant for its intended surgical application.
  Arms: OrACELL
Device: Connective Tissue Graft — A measured layer of dermis is surgically removed from the palate for use as a graft to cover gingival recession
  Other Names: Subepithelial Connective Tissue Graft
  Arms: Connective Tissue Graft

SUMMARY:
The purpose was to compare root coverage outcomes between autogenous connective tissue graft (CTG) and decellularized human dermis (OrACELL™) in areas of facial gingival recession.

DETAILED DESCRIPTION:
Twenty-four non-smoking, healthy patients, with 2mm or greater facial gingival recession at a minimum of one site that classified as a Miller Class I, II, or III recession defect were included. Patients were randomly assigned to either control (CTG) or OrACELL™ (test) groups, which were treated with identical surgical techniques. All root coverage clinical parameters were evaluated at baseline, 3-, and 6-months.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be between 18 and 80 years old, with recession present in one quadrant as either single or multiple buccal vertical recession sites
2. The defect must be at least 2mm in length, (measured from the CEJ to the midfacial gingival margin) and classified as either Miller Class I, II or III
3. Study is limited to vital and nonvital incisors, canines, and premolars
4. If teeth adjacent to the site to be treated had recession as well, they were included in the grafting procedure but not included in measurement
5. Plaque control defined as modified O'Leary Index of 85% was established before surgical intervention
6. Only sites with probing depths of 3mm or less and no bleeding on probing were accepted for surgery

Exclusion Criteria:

1. Subjects who smoke more than ten cigarettes per day or use nicotine replacement therapy
2. History of previous history of surgery performed at surgical sites included in study
3. Subjects who have uncontrolled or poorly controlled systemic conditions that could compromise or contraindicate periodontal surgery
4. Non-English speakers
5. Pregnant or lactating females
6. Immunosuppressant medications

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-03-26 (Actual); Primary Completion 2016-06-13 (Actual); Study Completion 2016-12-16 (Actual)

PRIMARY OUTCOMES:
Gingival Recession (Root Coverage) | 6 months
  The measurement in millimeters of the relationship of the cementoenamel junction (CEJ) to the gingival margin

IPD SHARING:
Plan to Share IPD: No